CLINICAL TRIAL: NCT01198288
Title: Randomised Controlled Trial on the Effects of Home-based Pulmonary Rehabilitation in Patients With Severe or Very Severe COPD
Brief Title: Effects of Home-based Pulmonary Rehabilitation in Patients With Severe or Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Riabilitatori Insufficienza Respiratoria (Other)
Responsible Party: Principal Investigator, Marta Lazzeri, Dr, Associazione Riabilitatori Insufficienza Respiratoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2010-09-07; First posted 2010-09-10 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Respiratory Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Drugs for COPD (as prescribed), oxygen therapy if needed*, check-up by the general practitioner and/or respirologist as usual.
  Educational leaflet regarding optimization of oxygen therapy and drugs; Benefits of physical activity and proposal of a programme of exercise training; Energy conservation techniques; Nutritional counselling; Activity of daily Living (ADL) diary; Prevention and management of acute exacerbation
  Monthly phone call with the aim of verifying:
  * the patients' clinical conditions;
  * the patient's adherence to the pharmacological treatments prescribed
  * the patient's compliance in filling out the clinical diary and the ADL diary
  Interventions: Other: Standard Care
- domiciliary rehabilitation (Experimental): Same as the standard care group plus 10 (ten) home-based visits supervised by a specifically trained respiratory therapist (education+exercise training) Autonomous home-based programme: The patients will be given instructions and training in order to continue the exercise training programme on the days the respiratory therapist is not visiting them.
  Counselling addressed at the outdoor activities.
  Interventions: Other: domiciliary rehabilitation

INTERVENTIONS:
Other: domiciliary rehabilitation — a respiratory rehabilitation programme at the patient home
  Arms: domiciliary rehabilitation
Other: Standard Care — As describe in the standard care arm
  Arms: Standard Care

SUMMARY:
This study will investigate if adding a domiciliary respiratory physiotherapy treatment to standard care in patients with chronic obstructive pulmonary disease (COPD) can improve physical function (walking test) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD (FEV1/FVC < 70% and FEV1 < 50% pred.) associated to hypoxaemic chronic respiratory insufficiency (PaO2 < 60mmHg) or
* Very severe COPD (FEV1/FVC < 70% and FEV1 < 30% pred.)

With the following characteristics:

* no signs of lung restriction (TLC≥80%)
* clinically stable for at least the last four weeks
* MRC ≥ 2
* no participation to PR programmes in the last year

FEV1= Forced expiratory volume in the 1st second FVC= Forced vital capacity TLC= Total Lung Capacity PaO2= Partial pressure of arterial oxygen

Exclusion Criteria:

* - Muscular-skeletal impairment that could limit the patient's participation to the exercise programme;
* Cognitive impairment that could limit the patient's participation to the activities of education and exercise, as assessed by the Mini Mental State (MMS) test <26;
* Malignancies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
meters as per walking test performance | 8 weeks

SECONDARY OUTCOMES:
Quality of life | 8 weeks
Bode index | 8 weeks
  This index is a combination of walking test result, Body Mass Index and respiratory measurement
dyspnea | 8 weeks
relapses | 8 weeks
services utilization | 8 weeks
  visits to the GP or Pneumologist that were not planned, hospital visits (emergency room )
meters as per walking test performance | 6 months
Quality of life | 6 months
Bode index | 6 months
  This index is a combination of walking test result, Body Mass Index and respiratory measurement
dyspnea | 6 months
relapses | 6 months
services utilization | 6 months
  visits to the GP or Pneumologist that were not planned, hospital visits (emergency room )
meters as per walking test performance | 12 months
Quality of life | 12 months
Bode index | 12 months
  This index is a combination of walking test result, Body Mass Index and respiratory measurement
dyspnea | 12 months
relapses | 12 months
services utilization | 12 months
  visits to the GP or Pneumologist that were not planned, hospital visits (emergency room )

CONTACTS AND LOCATIONS:
Locations (1):
- Unità di pneunologia, Ospedale di Busto Arsizio, Busto Arsizio, Varese, Italy